CLINICAL TRIAL: NCT03897556
Title: The Effect of High-Dose Guaraná on Cancer-Related Fatigue in Cancer Survivors
Brief Title: Effect of High-Dose Guarana And Cancer-Related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Luke Peppone, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3607
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Cancer-related Fatigue

STUDY DESIGN:
Intervention Model Description: This is a three-arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose (Active Comparator): This arm consists of cancer survivors who receive two guarana energy bars to take per day for six weeks; one in the morning and one around lunch time.
  Interventions: Dietary Supplement: Guarana herb
- Low-Dose (Active Comparator): This arm consists of cancer survivors who receive one guarana energy bar to take per day for six weeks; one in the morning only.
  Interventions: Dietary Supplement: Guarana herb
- Usual Care (Other): This arm receives usual-care only as cancer survivors.
  Interventions: Other: Usual Care

INTERVENTIONS:
Dietary Supplement: Guarana herb — The intervention is a functional food bar produced in a licensed commercial kitchen that contains guarana powder as well as dates, raisins, oats, spirulina, walnuts, flour, coconut butter, soybean oil, xanthan gum and chocolate chips.
  Arms: High-dose; Low-Dose
Other: Usual Care — Participant will receive 'usual-care' for cancer survivors. At the end of the study, after completing the Final Visit, they will receive 21 guarana energy bars to thank them for being in the study.
  Arms: Usual Care

SUMMARY:
This research will examine the effectiveness of a guaraná nutrition energy bar supplement on cancer-related fatigue based on scores from fatigue questionnaires. Participants will be randomized to one of three study arms: 1) two guaraná energy bars/day, 2) one guaraná energy bar/day 3) usual-care only/ no guaraná energy bars during study in cancer patients who have completed cancer treatment. We would also like to find out if this energy bar supplement improves physical performance, mood and reduces plasma glutamine and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of a malignant solid tumor between 4 and 36 months post-treatment (pathology report or MD documentation).
* Completed all forms of standard treatment (surgery, chemotherapy, radiation therapy, and/or immunotherapy) between 4 and 36 months prior to enrollment in the study.
* Be 18 years of age or older.
* Have cancer-related fatigue, as indicated by a response of a 4 or greater when asked to rate their level of fatigue at its worst in the past week on an 11-point scale anchored by "0": = 'no fatigue' and "10" = 'as bad as you can imagine' as taken from a single item question on the Symptom Inventory Questionnaire.
* Be able to read English (since the assessment materials are in printed format).

Exclusion Criteria:

* Participants must not: Have used guaraná supplements within the previous two months.
* Self-report that they are very sensitive to caffeine.
* Uncontrolled hypertension
* Have an allergy to walnuts, seaweed, soybeans and/or chocolate.
* Use medications for which caffeine intake is contraindicated including: β-adrenergic agonists, and/or medications that contain pseudoephedrine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
The change in mean level of cancer-related fatigue based on the Brief Fatigue Inventory survey | Baseline to final visit (six weeks)
  Participant will complete the Brief Fatigue Inventory Survey at baseline, midpoint and the final assessments. The scale is an 11-point scale, with a higher value indicating worse or greater level of fatigue.

SECONDARY OUTCOMES:
The adherence to taking guarana energy bars: participant ate ≥ 80% of the guaraná energy bars assigned to them over the course of the study. | Baseline to final visit (six weeks)
  Participants will bring in any leftover bars they don't consume during the study at midpoint and final assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmot Cancer Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
The information is not yet available to determine whether IPD should be made available to other researchers or not.